CLINICAL TRIAL: NCT05800834
Title: Effectiveness of Topical Morphine Use in Patients With Painful Neoplastic Wounds in the Breast and Head and Neck: Double Blind Randomized Clinical Trial - MorphineGEL
Brief Title: Benefits of Morphine Gel for Pain Reduction in Patients With Cancer Wounds
Acronym: MorphineGEL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Daianny Arrais de Oliveira da Cunha, Principal Investigator, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56160922.7.3001.5274
Record Dates: First submitted 2023-03-20; First posted 2023-04-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Wounds and Injuries; Cancer Pain; Cancer, Breast; Cancer Head Neck
Keywords: Malignant fungating wounds; Painful wounds; Palliative care
MeSH Terms: conditions — Wounds and Injuries; Cancer Pain; Breast Neoplasms; Head and Neck Neoplasms | interventions — Morphine; Lidocaine; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine sulfate (Experimental): Topical morphine with hydrogel base.
  Interventions: Drug: Morphine Sulfate
- Lidocaine Hcl 2% jelly (Active Comparator): 2% lidocaine jelly
  Interventions: Drug: Lidocaine Hcl 2% Jelly

INTERVENTIONS:
Drug: Morphine Sulfate — For the preparation of the gel formulated for the intervention, the proportion of an ampoule of dimorf® (morphine sulfate) in the injectable presentation of 10mg/ml will be used. Morphine sulfate is a strong, systemic opioid analgesic used for the relief of severe pain.
  For the base of the compound, Curatec Hidrogel with Alginate® will be used. A transparent and viscous hydrogel, which provides a moist environment, preventing the dressing from adhering to the skin, preventing additional injuries generated by difficulty removing the dressing.
  Other Names: Dimorf
  Arms: Morphine sulfate
Drug: Lidocaine Hcl 2% Jelly — The control group will receive lidocaine® in gel (2% sterile jelly lidocaine hydrochloride) alone. Because it is a homogeneous, transparent gel, free of lumps and impurities, it has similar characteristics to the hydrogel (Curatec Hidrogel with Alginate®) used in the preparation of morphine gel, guaranteeing the blinding of the study.
  Other Names: Lidocaine gel
  Arms: Lidocaine Hcl 2% jelly

SUMMARY:
The goal of this clinical trial is to compare in compare pain reduction in patients with malignant wounds using morphine gel or lidocaine gel. The main question to be answered is:

• Does morphine gel offer better pain control in malignant wounds when compared to lidocaine gel? Participants will answer a questionnaire where they report a note for pain at the site of the malignant wound and then the dressing will be performed by a nurse from the research team. The patient and the nurse do not know which product is being used. At the end of the dressing, the patient answers a new questionnaire. This process will be carried out for 3 days.

The researchers will compare the intervention group (morphine gel) and the control group (lidocaine gel) and verify if there is a difference in pain reduction between the two products.

DETAILED DESCRIPTION:
Potential participants will be all patients with malignant wounds in the head and neck or breast region who meet the inclusion and exclusion criteria, forming the study population.

After signing the free and informed consent form, the intervention group will receive topical morphine based on hydrogel in the formulation of 10mg of morphine sulfate - intravenous solution (1 ml) with 8g of hydrogel and the control group will receive lidocaine in gel.

To ensure the quality and accuracy of the data, in addition to the safety of the research participants, face-to-face monitoring visits will be carried out by the team from the Representative Area of Clinical Research (ARPC)/INCA throughout the execution of this protocol.

After signing the TCLE by the patient and researcher, the completion of the clinical form will begin. The pharmacist of the research team responsible for the randomization will be contacted to inform the inclusion of the patient in the study. The research team doctor will be responsible for prescribing the medication to be used, be it morphine or lidocaine gel, with a view to release by the hospital pharmacy.

Both morphine gel and lidocaine gel will be prepared in a flow hood suitable for handling the medications.

Adverse events will be reported, using medical terminology, in the source document and in the eCRF (electronic case report form). Upon identification of a reaction, the participant will be evaluated by the research team physician. All measures required for the treatment of the adverse event will be recorded in the source document.

Randomization and allocation will be performed using Research Electronic Data Capture (REDCap) software in a form that will only be viewed by non-blind members of the pharmacy team, responsible for handling the products and sending them to the team nurse who will be responsible for wound dressing evil.

The data collection forms (eCRF) will be customized in the REDCap software by the representative research area (ARPC) data management team. The data will be entered into the eCRFs according to the standard operating procedures of the Division of Clinical Research-INCA. The data will be exported to the R software by API (Application Programming Interface) where the statistical analyzes will be performed.

The sample size of each group was determined using the G*Power application (version 3.1.9.4), using the Wilcoxon and Mann-Whitney nonparametric test approach. The calculation suggests a minimum sample size of 53 patients per group.

In the first part of the analysis, a descriptive analysis of the sample profile and comparison of the baseline variables of the control and intervention groups will be performed. The second part will evaluate the effect of the treatments in the control and intervention groups, analyzing the significance of the observed differences and the size of the treatment effect.

For qualitative variables, the significance of the association between two variables, or the difference between the distribution of the proportions of the two groups, will be investigated using the chi-square test and, when it proves to be inconclusive, Fisher's exact test will be used.

The odds ratio (OR) will be the measure used to express some risk of a qualitative outcome when comparing the occurrence of the outcome in the groups.

For quantitative variables, the normality of distributions will be verified by the Kolmogorov-Smirnov and Shapiro-Wilk tests. If the variable of interest has a normal distribution in both groups, the comparison will be made using the student's t-test; if at least one of the groups does not present normal distribution, or if the variable to be compared is an ordinal scale, such as the pain scale, the comparison of the two groups will be performed using the Mann-Whitney test.

Two repeated measures in different evaluations will be compared by the paired Student's t-test, if the two measures present normal distribution, or by the Wilcoxon signed rank test, if at least one of the measures does not present normal distribution or if it is a scale measure ordinal.

More than two repeated measures will be compared by ANOVA for repeated measures, in the case of normality for all measures, or by the Friedman test, if at least one of the measures does not present normal distribution, or if it is an ordinal scale measure.

Classifications or qualitative factors observed repeatedly at different times will be compared by McNemmar test.

The effect of the received intervention on the pain score will be evaluated by the Glass effect size measure.

ELIGIBILITY:
Inclusion Criteria:

* Malignant neoplastic wound in breast or head and neck;
* Malignant neoplastic wound with staging >= II;
* KPS >=30%
* Having at least 3 on the numerical pain rating scale (0-10);
* Admission time equal to or greater than 48 hours.
* Make use of systemic morphine.

Exclusion Criteria:

* Wound with fistula;
* Wound with extensive coagulation necrosis (>50% of wound area;
* Exuding wound > 1 (PUSH Scale);
* Bleeding wound >1 (VIBe Scale)
* Ongoing radiotherapy on the wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 3 days
  The scale assesses the intensity of pain, where 0 means no pain and 10 means the most intense pain possible

SECONDARY OUTCOMES:
Pain relief | 3 days
  Difference in the means of pain assessed by the numeric pain assessment scale before and after the intervention.
General Comfort Questionnaire | 3 days
  General comfort questionnaire with scores ranging from 48-192, where 48 reports the worst comfort measure and 192 the highest comfort level reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Daianny A de Oliveira da Cunha, MSc., Principal Investigator — INCA Brazil
Locations (1):
- National Cancer Institute, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No